CLINICAL TRIAL: NCT00579085
Title: Double Blind Placebo Controlled Study of Outpatient Intravenous Ketamine for the Treatment of CRPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drexel University College of Medicine (Other)
Responsible Party: Dr. Robert J. Schwartzman MD, Drexel University College of Medicine
Organization: Drexel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16078-2-1 version 2
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Complex Regional Pain Syndrome
MeSH Terms: conditions — Complex Regional Pain Syndromes | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Other: IV NSS; Other: Normal Saline
- 2 (Experimental): INFUSION PLAN:
  All patients will be infused intravenously with 100 ml of normal saline with or without ketamine for four hours (25 ml/hr) daily for 10 days. The maximum intravenous ketamine infusion dose for this study will be 0.35 mg/kg/hr, not to exceed 25 mg/hr (100 mg of ketamine over a 4 hour period). On the first day, the intravenous ketamine infusion will be set to 50% of the maximum rate. On the second day, the intravenous ketamine infusion will be increased to 75% of the maximum rate. On the third day, the intravenous ketamine infusion will be increased to the maximum rate. The daily ketamine infusion rate is maintained at this level for the duration of the ten day study.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — IV Ketamine .35mg/kg times ten days.
  Arms: 2
Other: IV NSS — Placebo inactive ingredients
  Arms: 1
Other: Normal Saline — INFUSION PLAN:
  All patients will be infused intravenously with 100 ml of normal saline for four hours (25 ml/hr) daily for 10 days.Both patient arms will receive 2mg of Versed x two doses IV. They will also receive Clonidine (0.1 mg, po)
  Arms: 1

SUMMARY:
Complex Regional Pain Syndrome is a debilitating and extremely difficult to treat condition. There is a large body of evidence demonstrating the therapeutic value of N-methyl-D-aspartate (NMDA)-receptor antagonists in CRPS. The NMDA antagonist ketamine has been shown to be effective in the treatment of CRPS, resulting in complete remission of the disease in some patients. The purpose of this study is to evaluate intravenous outpatient infusion of sub-anesthetic doses of ketamine for the treatment of CRPS. A thorough evaluation of this procedure, providing information into the degree of relief and which of the constellation of RSD symptoms are best alleviated by this procedure would result in the optimization of this therapy for the treatment of CRPS.

DETAILED DESCRIPTION:
PRE TREATMENT:

Prior to treatment, after informed consent is obtained, each subject will be randomized into the ketamine or placebo (normal saline) infusion group. Both the patient and all other individuals involved in the study will be blinded as to the treatment except Guillermo Alexander PhD who will be responsible for the randomization and Margaret Rose RN who will be responsible for preparing the infusion solution. The patient will then receive a complete neurological examination and will be asked to complete a short form McGill and Quality of life questionnaires (Attachment 1).

Two weeks before treatment, 2 week and 3 months post treatment the following sensory and motor tests will be performed.

Thermal Detection Thresholds: Cool detection thresholds, which are mediated via A fibers and warm detection thresholds, which are mediated by small unmyelinated C fibers, will be determined using the TSA-II NeuroSensory Analyzer (Medoc Advanced Medical Systems U.S., Minneapolis, MN). The device consists of a computer controlled thermoelectric probe with a surface area of 9 cm2 that is attached using a velcro strap to the area of skin to be tested (thenar eminence and hypothenar eminence in the hands and the dorsal foot). For each trial the thermal stimulator starts at the thermo-neutral baseline temperature of 32oC, and increases for warming thresholds, or decreases for cooling thresholds, linearly at a rate of 1oC per second, until the subject pushes a button that stops and records the temperature and returns the unit to baseline temperature. Three trials are averaged for cool and for warm threshold for each site tested.

Thermal Pain: Thermal pain tolerance will be determined at the same sites and using the same method described above for thermal detection thresholds. The only difference is that for thermal pain trials, the subject will be instructed to push the control button (which immediately resets the stimulator back to baseline temperature) when the thermal stimulus (cold or hot) becomes painful. The TSA-II hardware automatically resets if the temperature reaches -10oC (for cooling) or 50oC (for heating) and the control button has not been pushed. This temperature range has been determined to not cause damage to skin or underlying tissue.

Dynamic Mechano-allodynia: Dynamic mechano-allodynia will be determined by stroking the skin three times within 5 seconds at a rate of 5 cm/sec with a 2.5 cm wide standard foam paintbrush. Allodynia severity will be measured on the subject's response using a numerical rating scale. The subject reports both the amount of pain on a 0-10 scale (0: no pain; 10: worst pain ever experienced) and the extent to which the sensation spread.

Static Mechano-allodynia and Temporal Summation: Static mechano-allodynia and temporal summation will be determined by pin-prick with a standard safety pin once every three seconds for a total of 5 times. The subject will be instructed to report the level of pain on a 0-10 scale (0: no pain; 10: worst pain ever experienced) and the extent to which the sensation spread after each repetition. The test will stop if the subject reports unacceptable pain at any point during the test.

Deep pressure pain thresholds: Deep pressure pain thresholds will be determined with a pressure algometer (Wagner Instruments, Greenwich, CT) which is a hand held device with a 1cm2 rub¬ber tip capable of measuring applied pressures of 0-5 kg. The device is held at a 90o angle to the body surface being tested. The pressure is gradually increased by 1 kg/second until the subject reports that the stimulus is painful or a pressure of 4 kg/cm2 has been reached. In the upper extremity thresholds to pain will be determined at: 1)second costosternal joint; 2) acromioclavicular joint; 3) lateral epicondyle; 4) radial styloid; 5) ulnar styloid; 6) second metacarpal; 6) fifth metacarpal. In the lower extremity thresholds to pain will be determined at: 1) greater trochanter; 2) lateral femoral condyle; 3) tibial tubercle; 4) mid shin; 5) medial malleolus; 6) lateral malleolus; 7) first metatarsal; 8) fifth metatarsal.

Quantification of Motor Function (finger tap): Finger tap rate will be determined using a computer program developed by our group. The subject is instructed to press the spacebar of a standard computer keyboard as fast as possible with the index finger of each hand respectively for 30 seconds. The program determines the rate and plots the results.

Cutaneous Temperature: Skin temperature will be measured by use of an infra-red thermometer (Dermatemp Infrared Temperature Scanner, model DT-1001, Exergen Corp., Watertown, MA)

A pregnancy test will be administered to all females of child bearing potential and blood will also be drawn for SMA-20, CBC w/ Differential and a full thyroid panel. All subjects will be asked to wear an activity watch until the treatment begins (two week). This watch (Attachment 2) will evaluate the subject's level of activity and at random programmed intervals records the subject's pain level for the two weeks prior to treatment. This is accomplished by sounding a tone at which time the subject is instructed to presses a key pad and enter a number from 0-10 (0 = no pain and 10 = unbearable pain). The patient will be asked to complete the short form McGill and Quality of life questionnaires weekly until the start of the infusions.

PRE INFUSION:

On the first day of treatment but prior to the start of the infusions, the patient will be weighed, undergo a neurologic exam, have vital signs evaluated and have an intravenous line inserted.

On all ten treatment days, patients on both the ketamine and placebo groups are placed on the cardiac monitor for cardiac rhythm, blood pressure, pulse and oxygen saturation monitoring. In addition, Clonidine (0.1 mg, po) and Versed (4 mg, iv) will be administered. Clonidine has been shown, in animals, to potentiate the neuropathic pain-relieving action of NMDA receptor blockers like ketamine while preventing their neurotoxic side effects. Versed at this dose, provides mild sedation and relieves anxiety.

INFUSION PLAN:

All patients will be infused intravenously with 100 ml of normal saline with or without ketamine for four hours (25 ml/hr) daily for 10 days. The maximum intravenous ketamine infusion dose for this study will be 0.35 mg/kg/hr, not to exceed 25 mg/hr (100 mg of ketamine over a 4 hour period). On the first day, the intravenous ketamine infusion will be set to 50% of the maximum rate. On the second day, the intravenous ketamine infusion will be increased to 75% of the maximum rate. On the third day, the intravenous ketamine infusion will be increased to the maximum rate. The daily ketamine infusion rate is maintained at this level for the duration of the ten day study.

CONSIDERATIONS: (Other Treatments and Meds)

Increased salivation:

Glycopyrrolate (Robinul) Initially 1mg TID then maintenance dose BID prn

Psychiatric symptoms:

Ativan 1mg - HAVE AVAILABLE prn Continued use of current medications with the exception of NMDA receptor blockers such as amantadine, memantine, Magnesium sulfate.

Administer other adjuncts prn O2 2-3 L/min. via Nasal Cannula - HAVE AVAILABLE prn

LABS:

Ketamine Level (red top tube) on infusion days 1, 5, 6 and 10.

NURSING CARE & ORDERS:

During the IV Ketamine Infusion:

Continuous cardiac monitoring, Pulse oximetry with q 1 hr blood pressure monitoring V/S q 1 hr Versed (2 mg iv) administration may be repeated two hours into or at the completion of the infusion.

Activity:

Patient can leave infusion chair with assistance for bathroom visit. Patient is allowed to bring head set (music) or a book to read. No cell phones or laptop computers are allowed.

Following the last (10th) infusion, the patient will be seen at two weeks then monthly at the Neurology Pain Clinic for the following 3 months. All subjects will be asked to wear an activity watch from the time of the last infusion until the two week post treatment visit. Patients will be instructed to complete the

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CRPS based on the modified IASP (International Association for the Study of Pain) research criteria (Harden RN and Bruehl SP
* Diagnostic Criteria: The Statistical Derivation of the Four Criterion Factors.
* In CRPS: Current Diagnosis and Therapy, Progress in Pain Research and Management, Vol 32: pp 45-58, 2005), whose condition is intractable for at least six months and have failed at least three of the following therapies:

  * Nerve blocks
  * Opioid analgesics
  * Non-opioid analgesics
  * Non-steroidal anti-inflammatory drugs
  * Anti-seizure medications
  * Antidepressants
  * Muscle relaxants; or
  * Physical therapy.
* The patients must be ketamine naïve and can be of either gender including all racial and minority groups. The patient's age must be between 18 and 65 years, inclusive.
* The study subjects must report pain levels equal to or greater than 4 on a scale of 0-10 (0 = no pain and 10 = unbearable pain). The pain must be stable over time and not vary more that 1 pain level.
* The patient must be on a stable dose of CRPS medications for 28 days prior to and throughout the duration of the study.
* The patient must be accompanied by a responsible adult.
* The patient will be instructed that he/she will not be allowed to drive home following the infusion. Therefore in order to be included in the study the subjects must arrange for transportation for the 10 day duration of the study.

Exclusion Criteria:

* Patients less than 18 years of age will be excluded. In this initial study, patients over 65 years of age will be excluded due to possible unforeseen concomitant medical problem.
* Patients that have previously undergone intravenous ketamine infusions will be excluded from the study.
* Patients who are pregnant, are lactating, have known psychotic or psychiatric illness, are afflicted with glaucoma or have thyrotoxicosis will also be excluded.
* Any patient that is unable to provide consent due to cognitive difficulties will not be used in this study.
* Patients that can not provide the means to be transported home following daily infusions will be excluded from the study.
* The investigators feel that issues concerning monetary gain and or loss due to the patient's medical condition may adversely affect the study, therefore, patients with active litigation, compensation or disability issues related to their CRPS will be excluded.
* Patients with a history of substance abuse will be excluded.
* Patients on certain blood pressure lowering medications such as calcium blockers, or beta blockers will be excluded from the study.
* Patients with major medical problems including but not limited to; uncontrolled hypertension, hypotension, cardiac failure, renal failure or liver failure will not be used in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-09; Primary Completion 2008-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is to evaluate intravenous outpatient infusion of sub-anesthetic doses of ketamine for the treatment of CRPS by a 30% pain reduction post treatment | Patients will be evaluated for three months after treatment

SECONDARY OUTCOMES:
Lenght of relief of pain | When and if pain returns to pre treatment levels

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University College of Medicine Department of Neurology, Philadelphia, Pennsylvania, United States